CLINICAL TRIAL: NCT03061435
Title: Screening for Anal Cancer in Women With High-grade Vulvar Dysplasia or Vulvar Cancer.
Acronym: Vulvar-AIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Danielle Vicus (Other)
Responsible Party: Sponsor-Investigator, Dr. Danielle Vicus, Dr. Danielle Vicus, MD, MSc, FRCSC, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GYNEOCC 3
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Vulvar Cancer; Cervical Cancer; Vulvar Dysplasia; Cervical Dysplasia; Anal Cancer; Anal Dysplasia; HPV-Related Anal Squamous Cell Carcinoma
Keywords: Vulvar Cancer; Cervical Cancer; Vulvar Dysplasia; Cervical Dysplasia; Anal Cancer; Anal Dysplasia; HPV
MeSH Terms: conditions — Vulvar Neoplasms; Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Anus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Screening anal Pap Smear - Negative (75%) (Other): All patients will receive an anal Pap test. 75% of patients with a negative anal Pap will complete study with no further intervention.
  Interventions: Procedure: Screening anal Pap smear - No high-resolution anoscopy
- Screening anal Pap Smear - Negative (25%) (Other): All patients will receive an anal Pap test. Remaining 25% of patients will proceed to high-resolution anoscopy (HRA) clinic to assess the negative predictive rate of HRA.
  Interventions: Procedure: Screening anal Pap smear - High-resolution anoscopy
- Screening anal Pap Smear - Positive (Other): All patients will receive an anal Pap test. Any patient with abnormal cytology on their Pap test will be referred to HRA clinic for management. This includes potential biopsy and treatment.
  Interventions: Procedure: Screening anal Pap smear - High-resolution anoscopy

INTERVENTIONS:
Procedure: Screening anal Pap smear - No high-resolution anoscopy — 75% of patients with negative cytology on their anal Pap smear will not receive high-resolution anoscopy
  Arms: Screening anal Pap Smear - Negative (75%)
Procedure: Screening anal Pap smear - High-resolution anoscopy — 25% of patients with negative cytology on their anal Pap smear will receive high-resolution anoscopy. All patients with positive (abnormal) cytology on their anal Pap smear will receive high-resolution anoscopy.
  Arms: Screening anal Pap Smear - Negative (25%); Screening anal Pap Smear - Positive

SUMMARY:
Almost half of all women will develop an HPV infection in their lifetime. While most infections are naturally asymptomatic or cleared by the immune system, some persist and can lead to the development of cervical, vulvar, or anal lesions and eventually cancer. Screening regimens for these lesions are currently only in place for the cervix through regular Pap tests. These Pap tests usually involve an examination of the vulva -however, no screening procedures exist for anal cancer for women. Several studies have suggested that women with existing gynecological lesions are more likely to develop anal lesions and anal cancer. Here the investigators propose a multi-center study which seeks to screen for and treat anal cancer in women over the age of 40 with vulvar lesions and a stable immune system. The investigators will achieve this through performing anal Pap smears on eligible women and conducting High Resolution Anoscopy (HRA) and appropriate treatment procedures on those with abnormal anal cells. With enough evidence, there may be an indication to establish regular anal cancer screening measures in this potentially underserved population.

Hypothesis: The investigators hypothesize that at least 40% of women with vulvar cancer or VIN2/3 will have abnormal anal cytology. 35% of the population will be hrHPV DNA positive and 11% will additionally have AIN2/3. This prospective study may lay the groundwork for routine anal screening regimens in Ontario and help shift health policy to treat this population.

ELIGIBILITY:
Inclusion Criteria:

* Women age ≥ 40
* Previous diagnosis of VIN 2/3 or vulvar

Exclusion Criteria:

* Women with a previous diagnosis of cancer aside from basal cell carcinoma of the skin, cervical cancer, or vulvar cancer
* Women who are HIV positive
* Women currently taking immunosuppressant medication
* Women who have had a previous hysterectomy

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of abnormal anal cytology and hrHPV DNA in women with VIN 2/3 or vulvar cancer | 6 months to 1 year

SECONDARY OUTCOMES:
Prevalence of AIN in women with VIN 2/3 or vulvar cancer | 6 months to 1 year
Assess t he correlation between abnormal anal cytology, hrHPV DNA, and AIN | 6 months to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Vicus, MD, Principal Investigator — Odette Cancer Centre
Locations (1):
- Odette Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No